CLINICAL TRIAL: NCT05960383
Title: Comparison Between Rapid Molecular Technique BioFire Pneumonia Panel Filmarray and Conventional Culture-based Methods in the Microbiologic Diagnosis on Bronchoalveolar Lavage Fluid of Lung Transplant Patients
Brief Title: Molecular vs Conventional Microbiologic Diagnosis for Infections in Lung Transplantation
Acronym: PNEUMOARRAY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 665_2022bis
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Lung Transplant Infection; Molecular Diagnostic; Bacterial Infections; Pneumonia; Tracheobronchitis
Keywords: Lung transplant; Infection
MeSH Terms: conditions — Bacterial Infections; Pneumonia; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Lung transplant patients: 53 patients who receive lung transplant and undergo microbiologic assessment with BioFire Pneumonia Panel Plus and conventional culture
  Interventions: Diagnostic Test: BioFire Pneumonia Panel Plus

INTERVENTIONS:
Diagnostic Test: BioFire Pneumonia Panel Plus — Assessment of sensbility and specificity of BioFire Pneumonia Panel Plus in lung transplantation

SUMMARY:
The goal of this prospective study is to compare rapid molecular technique BioFire Pneumonia Panel Filmarray and conventional culture-based methods in the microbiologic diagnosis on bronchoalveolar lavage of lung transplant patients.

The main questions it aims to answer are:

* determine the microbiological concordance between molecular diagnostic and conventional culture techniques on donor's bronchoalveolar lavage before lung transplantation
* determine the microbiological concordance between molecular diagnostic and conventional culture techniques on recipient's bronchoalveolar lavage, performed 72 hours after lung transplantation
* determine the microbiological concordance between molecular diagnostic and conventional culture techniques in detecting molecular resistance patterns
* determine the difference in time to microbiological results between molecular diagnostic and conventional culture techniques
* determine time to clinical decision based on molecular diagnostic techniques compared to conventional culture techniques

DETAILED DESCRIPTION:
Molecular assays that detect bacterial organisms by nucleic acid sequences rather than culture have the potential to improve time to diagnosis for lower respiratory tract infections. However, their performance characteristics are unknown in lung transplant recipients.

PNEUMOARRAY is a prospective study, including all patients aged >18 years that undergo lung transplantation from September 2022, at IRCCS Fondazione Cà Granda Policlinico in Milan. Patients who do not meet inclusion criteria are excluded from this study.

A fibro-bronchoscopy (FBS) with bronchoalveolar lavage (BAL) is performed, according to clinical practice, both on lungs donor and recipient. Donor's BAL is collected before graft transplantation, while BAL on lung transplant recipient is performed 72 hours after transplantation. On each BAL sample, both of lung donor and recipient, molecular diagnostic and culture exam are performed.

The goal of this prospective study is to compare rapid molecular technique BioFire Pneumonia Panel Filamarray and conventional culture-based methods in the microbiological diagnosis on bronchoalveolar lavage of lung transplant patients.

The primary outcome is:

-determine the microbiological concordance between molecular diagnostic and conventional culture techniques on donor's bronchoalveolar lavage before lung transplantation

Secondary outcomes are:

* determine the microbiological concordance between molecular diagnostic and conventional culture techniques on recipient's bronchoalveolar lavage, performed 72 hours after lung transplantation
* determine the microbiological concordance between molecular diagnostic and conventional culture techniques in detecting molecular resistance patterns
* determine the difference in time to microbiological results between molecular diagnostic and conventional culture techniques
* determine time to clinical decision based on molecular diagnostic techniques compared to conventional culture techniques

Sample size for statistical significance includes 53 patients.

For the majority of bacteria and fungi, microbiological culture from BAL remains the gold standard for diagnosis, but cultures are limited by long turnaround time and decreased sensitivity in patients that have received empiric anti-infective therapy. In this setting, fast microbiological diagnosis may be crucial to begin targeted antimicrobial therapy/prophylaxis and identify genes encoding resistance, in order to administer targeted therapy and to reduce antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* all patients aged >18 years that undergo lung transplantation from February 2023, at IRCCS Fondazione Cà Granda Policlinico in Milan and performed FBS+BAL

Exclusion Criteria:

* Patients who do not meet inclusion criteria are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PNEUMOARRAY is a prospective study, including all patients aged >18 years that undergo lung transplantation from February 2023, at IRCCS Fondazione Cà Granda Policlinico in Milan. Patients who do not meet inclusion criteria are excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
microbiological concordance on donor's BAL | 2023-2024
  determine the microbiological concordance between molecular diagnostic and conventional culture techniques on donor's bronchoalveolar lavage before lung transplantation

SECONDARY OUTCOMES:
microbiological concordance on recipient's BAL | 2023-2024
  determine the microbiological concordance between molecular diagnostic and conventional culture techniques on recipient's bronchoalveolar lavage, performed 72 hours after lung transplantation
concordance in in detecting molecular resistance patterns | 2023-2024
  determine the microbiological concordance between molecular diagnostic and conventional culture techniques in detecting molecular resistance patterns
difference in time to microbiological results | 2023-2024
  determine the difference in time to microbiological results between molecular diagnostic and conventional culture techniques
determine time to clinical decision | 2023-2024
  determine time to clinical decision based on molecular diagnostic techniques compared to conventional culture techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Fondazione Ca' Granda Policlinico Di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR